CLINICAL TRIAL: NCT04766775
Title: The Pharmacokinetics of Silver Diamine Fluoride (SDF) in Healthy Children
Acronym: SDF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Dr Lim Siau Peng, Principal Investigator, Postgraduate student year 3, Department of Paediatric Dentistry, University of Malaya
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: DF CD1914/0065/20157 (P)
Record Dates: First submitted 2021-02-04; First posted 2021-02-23 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Dental Caries in Children
Keywords: silver diamine fluoride

STUDY DESIGN:
Intervention Model Description: ll of the patients enrolled in the study (aged 4 to 10 years old) will receive Silver Diamine Fluoride (SDF) treatment to the decayed primary tooth/teeth by having the application of Silver Diamine Fluoride (SDF) onto the tooth cavity. The weight of the SDF capsule and brush will be measured before and after the SDF application. This step approximates the amount of SDF applied to the tooth surface. Urine and hair samples will be taken to assess the silver and fluoride levels. Urine samples will be taken before the SDF treatment, in the first and second 24 hours after the SDF treatment. For the hair samples, it will be taken before the SDF treatment as well as day 7,14,30,60,75, and 90 after the SDF treatment. After the day 90 review, if caries remains active, the SDF treated teeth will be restored or undergo a six-monthly SDF application.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Application of Silver Diamine Fluoride onto the carious teeth surfaces (Other): The patients will receive Silver Diamine Fluoride (SDF) treatment to the carious primary teeth. These are teeth with no sign or symptom, radiographically the deepest layer of the caries lesion does not involve the pulp, the inter-radicular area appears normal). Procedure: apply vaseline, isolate the tooth with a cotton roll, remove the food debris, and gross plaque on the tooth cavity with a spoon excavator, dry the tooth, apply the SDF (a clear, colorless solution) onto the tooth cavity. This application lasts for one minute. Take the urine and hair sample to assess the silver and fluoride levels. Take the urine sample before the SDF treatment, in the first and second 24 hours after the SDF treatment. Take the hair samples before the SDF treatment, followed by days 7,14,30,60,75, and 90 after the SDF treatment. Send the hair and urine samples to the laboratory to assess the silver and fluoride levels. If caries remains active, restore the SDF treated after the day 90 review.
  Interventions: Device: Silver Diamine Fluoride

INTERVENTIONS:
Device: Silver Diamine Fluoride — Silver Diamine Fluoride (Riva Star) which contains silver, fluoride, ammonia and water.

SUMMARY:
This study focus on the pharmacokinetic characteristic of silver diamine fluoride (SDF) in healthy children. All of the children received treatment for the decayed teeth in the same way. A medication called silver diamine fluoride is used to treat the decayed teeth. It contains a high concentration of fluoride (range from 14100 ppm to 51013 ppm) and silver. This medication halts the decay process through the combined effects of anti-bacterial from silver and remineralization from fluoride. As this product contains the highest concentration of fluoride level found in the market and the metal element of silver, the investigators aim to study the body's reaction towards SDF. The investigators collect the hair and urine samples at different time points and then analyze them to determine the silver and/or fluoride levels. The outcomes include 1. the silver level in the hair and urine samples 2. the fluoride level in the urine samples. The investigators analyze the silver level in hair and urine samples using Inductively Coupled Plasma Mass Spectrometry (ICP-MS); fluoride level in urine samples using Ion-Selective Electrode.

DETAILED DESCRIPTION:
This research aims to determine the pharmacokinetics characteristics of silver and fluoride following topical application of Silver Diamine Fluoride (SDF) in healthy children. The use of Silver Diamine Fluoride is increasingly widespread since the device is approved by the Food and Drug Administration (FDA) of the United States in 2014, especially among the pediatric population. It is a single-arm, clinical study with the specific objectives: 1. to assess the level of silver and fluoride in the urine sample of patients receiving the SDF treatment; 2. to evaluate the pharmacokinetics of silver, based on the hair sample of patients receiving the SDF treatment. The investigators hypothesize that the pharmacokinetic characteristics of silver diamine fluoride in healthy children are different from that of silver diamine fluoride in healthy adults. The research is taking place at the Paediatrics Dentistry Specialist Clinic, Faculty of Dentistry, University of Malaya. The investigators have used a convenience sampling method to recruit children aged 4-10 years old to join the study. The investigators have calculated the sample size based on the alpha error probability of 0.05 and the power of study at 95%. The investigators have recruited children with at least one decayed primary tooth without clinical signs or symptoms. Radiographically the deepest layer of caries lesion does not involve the pulp. The investigators have excluded children with known medical illness, having glass ionomer or stainless steel crown restorations in the oral cavity. All of the recruited patients received the same intervention, the application of SDF onto the tooth cavity. The investigators have taken the patients' biological samples (urine and hair) to assess the silver and/or fluoride levels. The urine samples are collected before the SDF treatment, in the first and second 24 hours after the SDF treatment. Besides that, hair samples are collected before the SDF treatment, followed by days 7,14,30,60,75, and 90 after the SDF treatment. The silver level in hair and urine samples were analyzed using Inductively Coupled Plasma Mass Spectrometry (ICP-MS); fluoride level in urine samples using Ion-Selective Electrode. After review at days 90, if caries remains active despite the SDF treatment, the investigators will restore the SDF treated teeth or continue the six-monthly application of SDF depending on the patient's ability to cope with the procedure and the caries status.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy children aged between 4 to 10 years old

* With at least one decayed primary tooth without clinical signs or symptoms suggesting reversible or irreversible pulpitis.
* Radiographically the deepest layer of caries lesion does not encroach on pulp, and inter-radicular supporting structures appear normal

Exclusion Criteria:

1. Children aged below 4 years and above 10 years
2. Healthy children aged between 4 to 10 years old

   * Do not have decayed teeth
   * The decayed tooth with clinical signs or symptoms suggesting reversible or irreversible pulpitis
   * Radiographically the deepest layer of caries lesion does encroach on pulp, and inter-radicular supporting structures appear abnormal
   * No consent and permission to join the study
   * Taking medications/over the counter medications/supplements
   * Known allergy to silver or fluoride
   * Presence of ulcer in the mouth which has not heal completely
   * Presence of at least one tooth treated with silver fillings or stainless steel crown.
   * Presence of at least one tooth filled with a material that contains glass particles known as glass ionomer within a year before this research.
   * Children with medical problems

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2020-07-03 (Actual); Primary Completion 2020-11-26 (Actual); Study Completion 2021-11-26 (Estimated)

PRIMARY OUTCOMES:
To assess the silver level in the hair samples (µg/g) | 7 days
  SDF treatment will be provided to the patients, hair samples will be collected at day 7 after the SDF treatment
To assess the silver level in the hair samples (µg/g) | 14 days
  SDF treatment will be provided to the patients, hair samples will be collected at day 14 after the SDF treatment
To assess the silver level in the hair samples (µg/g) | 30 days
  SDF treatment will be provided to the patients, hair samples will be collected at day 30 after the SDF treatment
To assess the silver level in the hair samples (µg/g) | 60 days
  SDF treatment will be provided to the patients, hair samples will be collected at day 60 after the SDF treatment
To assess the silver level in the hair samples (µg/g) | 75 days
  SDF treatment will be provided to the patients, hair samples will be collected at day 75 after the SDF treatment
To assess the silver level in the hair samples (µg/g) | 90 days
  SDF treatment will be provided to the patients, hair samples will be collected at day 90 after the SDF treatment
To assess the fluoride level in the urine samples (µg/24h) | 72 hours
  SDF treatment will be provided to the patients, urine samples will be collected before the start of the treatment; in the first and second 24 hour after the treatment
To assess the silver level in the urine samples (µg/24h) | 72 hours
  SDF treatment will be provided to the patients, urine samples will be collected before the start of the treatment; in the first and second 24 hour after the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Siau Peng Lim, DDS (USM), Principal Investigator — University of Malaya, Faculty of Dentistry
Locations (1):
- University of Malaya, Kuala Lumpur, Kuala, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vasquez E, Zegarra G, Chirinos E, Castillo JL, Taves DR, Watson GE, Dills R, Mancl LL, Milgrom P. Short term serum pharmacokinetics of diammine silver fluoride after oral application. BMC Oral Health. 2012 Dec 31;12:60. doi: 10.1186/1472-6831-12-60. PMID 23272643
- [Background] Chen KF, Milgrom P, Lin YS. Silver Diamine Fluoride in Children Using Physiologically Based PK Modeling. J Dent Res. 2020 Jul;99(8):907-913. doi: 10.1177/0022034520917368. Epub 2020 May 6. PMID 32374712
- [Background] Lansdown AB. Silver in health care: antimicrobial effects and safety in use. Curr Probl Dermatol. 2006;33:17-34. doi: 10.1159/000093928. PMID 16766878
- [Background] Crystal YO, Marghalani AA, Ureles SD, Wright JT, Sulyanto R, Divaris K, Fontana M, Graham L. Use of Silver Diamine Fluoride for Dental Caries Management in Children and Adolescents, Including Those with Special Health Care Needs. Pediatr Dent. 2017 Sep 15;39(5):135-145. PMID 29070149
- [Background] Lansdown AB. Silver. I: Its antibacterial properties and mechanism of action. J Wound Care. 2002 Apr;11(4):125-30. doi: 10.12968/jowc.2002.11.4.26389. PMID 11998592
- [Background] Ngara B, Zvada S, Chawana TD, Stray-Pedersen B, Nhachi CFB, Rusakaniko S. A population pharmacokinetic model is beneficial in quantifying hair concentrations of ritonavir-boosted atazanavir: a study of HIV-infected Zimbabwean adolescents. BMC Pharmacol Toxicol. 2020 Aug 3;21(1):58. doi: 10.1186/s40360-020-00437-y. PMID 32746923
- [Background] Cooper GA, Kronstrand R, Kintz P; Society of Hair Testing. Society of Hair Testing guidelines for drug testing in hair. Forensic Sci Int. 2012 May 10;218(1-3):20-4. doi: 10.1016/j.forsciint.2011.10.024. Epub 2011 Nov 15. PMID 22088946
- [Background] Kintz P. Hair Analysis in Forensic Toxicology: An Updated Review with a Special Focus on Pitfalls. Curr Pharm Des. 2017;23(36):5480-5486. doi: 10.2174/1381612823666170929155628. PMID 28969544
- [Result] Lin YS, Rothen ML, Milgrom P. Pharmacokinetics of 38% topical silver diamine fluoride in healthy adult volunteers. J Am Dent Assoc. 2019 Mar;150(3):186-192. doi: 10.1016/j.adaj.2018.10.018. PMID 30803490
- [Result] Villa A, Anabalon M, Zohouri V, Maguire A, Franco AM, Rugg-Gunn A. Relationships between fluoride intake, urinary fluoride excretion and fluoride retention in children and adults: an analysis of available data. Caries Res. 2010;44(1):60-8. doi: 10.1159/000279325. Epub 2010 Feb 2. PMID 20130402
- [Result] Wilschefski SC, Baxter MR. Inductively Coupled Plasma Mass Spectrometry: Introduction to Analytical Aspects. Clin Biochem Rev. 2019 Aug;40(3):115-133. doi: 10.33176/AACB-19-00024. PMID 31530963
- [Result] DiVincenzo GD, Giordano CJ, Schriever LS. Biologic monitoring of workers exposed to silver. Int Arch Occup Environ Health. 1985;56(3):207-15. doi: 10.1007/BF00396598. PMID 4066049
- [Result] Goulle JP, Mahieu L, Castermant J, Neveu N, Bonneau L, Laine G, Bouige D, Lacroix C. Metal and metalloid multi-elementary ICP-MS validation in whole blood, plasma, urine and hair. Reference values. Forensic Sci Int. 2005 Oct 4;153(1):39-44. doi: 10.1016/j.forsciint.2005.04.020. PMID 15979835
- [Result] World Health Organization. (2014). Basic methods for assessing renal fluoride excretion in community prevention programmes for oral health. World Health Organization. https://apps.who.int/iris/handle/10665/112662

DOCUMENTS (1):
  • Informed Consent Form (2020-07-01): https://cdn.clinicaltrials.gov/large-docs/75/NCT04766775/ICF_000.pdf